CLINICAL TRIAL: NCT01534130
Title: Acupuncture for the Sleep Disorder of Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Principal Investigator, Li ying, Principal Investigator, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30801488
Record Dates: First submitted 2011-12-14; First posted 2012-02-16 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome; Sleep Disorder, Adjustment; Acupuncture
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Dyssomnias | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental)
  Interventions: Device: Acupuncture
- sham acupuncture (Sham Comparator)
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — Participants will receive five sessions of verum acupuncture in the first week after randomization, three sessions in the second and third weeks after randomization, and two sessions in the forth week after randomization.
  Other Names: Streitberger needles(Special No.16)
  Arms: acupuncture
Device: Sham acupuncture — Participants will receive five sessions of sham acupuncture in the first week after randomization, three sessions in the second and third weeks after randomization, and two sessions in the forth week after randomization.
  Other Names: Streitberger Placeboneedles(Gauge 8 x 1.2"/0.30 x 30 mm).
  Arms: sham acupuncture

SUMMARY:
The investigators will conduct acupuncture for participants with chronic fatigue syndrome(CFS). Firstly the investigators aim to figure out the characteristic of sleep structure of CFS and the changes caused by acupuncture. Secondly the investigators seek to investigate the characteristic of sleep-wake rhythm, slow wave sleep(SWS)-rapid eye movement(REM)sleep rhythm, and REM sleep rhythm of CFS and the readjusting of acupuncture for it. Thirdly the investigators want to know the efficacy of acupuncture for relieving the fatigue, reducing accompanying symptoms and for improving the life quality of CFS.

DETAILED DESCRIPTION:
This trial is a randomized, placebo controlled clinical trial. 72 participants with CFS are randomly allocated to two different groups. Treatment group is acupuncture, while the control group is sham acupuncture. The ratio of treatment group and control group is 2:1. Both acupuncture and sham acupuncture group will receive 12 sessions of verum/sham acupuncture in 4 weeks.

The result of this trial (available in 2011) will supply evidence on the efficacy of acupuncture for sleep disorder of CFS.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who meet the diagnosis criteria of CFS;
2. Clinically evaluated, exclude any disease that can explain the chronic fatigue;
3. The onset age of CFS is between 18 and 50 years old;
4. Have not taken any hypnotic, melatonin, or antidepressants within 45 days;
5. Willing to finish the whole observation period;
6. With written consent form signed by themselves.

Exclusion Criteria:

1. Chronic fatigue caused by diseases such as internal diseases(for example, pulmonary emphysema, rheumatoid arthritis, etc.), mental illness(for example, any type of dementia paranoids, depression, etc.), some diseases that just onset or evaluated (for example, sleep deprivation, untreated diabetes, etc.), some diseases that need recovery gradually(for example, restless legs syndrome, lactation, etc.), morbid obesity;
2. Participants in other clinical research;
3. Pregnant women, lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The sleep perception | Change from baseline in sleep perception at 4 weeks
  The percentage of the ratio between the total sleep time perceived by the patient and the total sleep time obtained by PSG.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index(PSQI) | Change from baseline in PSQI at 4 weeks
The Fatigue Severity Scale(FSS) | Change from baseline in FSS at 4 weeks
The Somatic and Psychological Health Report(SPHR) | Change from baseline in SPHR at 4 weeks
The Medical outcomes Study 36-Item Short-Form Health Survey questionnaire(SF-36) | Change from baseline in SF-36 at 4 weeks
Sleep-wake rhythm | Change from baseline in sleep-wake rhythm at 4 weeks
DSWS-REM sleep rhythm | Change from baseline in DSWS-REM sleep rhythm at 4 weeks
REM sleep rhythm | Change from baseline in REM sleep rhythm at 4 weeks
Sleep latency | Change from baseline in sleep latency at 4 weeks
Total sleep time | Change from baseline in total sleep time at 4 weeks
Sleep efficiency | Change from baseline in sleep efficiency at 4 weeks
Percentage of every sleep stage | Change from baseline in percentage of every sleep stage at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, A.P., Study Director — School of Acupuncture& Tuina，Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu university of Traditonal Chinese Medcine, Chengdu, Sichuan, China